CLINICAL TRIAL: NCT04574024
Title: Effect of High-fiber Supplement in Multiple Sclerosis
Brief Title: HFS (High-Fiber Supplement) in MS (Multiple Sclerosis)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Suhayl Dhib-Jalbut, MD (Other)
Responsible Party: Sponsor-Investigator, Suhayl Dhib-Jalbut, MD, Professor of Neurology, Rutgers, The State University of New Jersey
Organization: Rutgers, The State University of New Jersey (Other)
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: Pro2019001677
Record Dates: First submitted 2020-09-21; First posted 2020-10-05 (Actual); Results first posted 2024-12-17 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-11

CONDITIONS: Multiple Sclerosis
Keywords: High-fiber supplement
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Intervention Model Description: High-fiber supplement-treatment and non-treatment
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MS study cohort (Other): Baseline: 7 MS patients enrolled for the study. No treatment or before treatment.
  NBT-NM108-Treatment for 8 weeks: 3 out of 7 MS patients consumed the NBT-NM108 for 8 weeks.
  NBT-NM108-Treatment for 12 weeks: 2 MS patients further consumed the NBT-NM108 for four more weeks.
  Patients consumed dietary fiber three times a day at 60 g/day
  Interventions: Drug: NBT-NM108

INTERVENTIONS:
Drug: NBT-NM108 — MS Patients received NBT-NM108 at 60 g/day.

SUMMARY:
Multiple sclerosis (MS) is an autoimmune disease directed against the Central Nervous System (CNS). Recent studies have indicated that changes in the gut microbiota are associated with disease initiation and progression. The reduction of bacterial taxa involved in producing health-promoting metabolites, such as short-chain fatty acids (SCFAs), has been reported in MS patients. SCFAs play an important role in the suppression of inflammation. The levels of SCFAs in the blood of MS patients are significantly reduced when compared to those of healthy controls. Since the intake of dietary fiber increases the growth of SCFA-producing bacteria, we investigated the effect of a high-fiber supplement (HFS) on gut bacteria and immunological parameters in MS patients.

DETAILED DESCRIPTION:
Our collaborator, Dr. Liping Zhao, developed a high-fiber supplement (HFS), NBT-NM108. His recent study has suggested an association between intake of NBT-NM108 and increased abundance of short-chain fatty acid (SCFA)-producing gut bacteria. Recent studies have suggested that Relapsing-Remitting Multiple Sclerosis (RRMS) is associated with gut dysbiosis, alteration of gut bacteria, and decreased production of SCFAs. Therefore, we have investigated the effect of NBT-NM108 on RRMS-associated gut dysbiosis and the cytokines produced by immune cells. Seven patients were enrolled, and their stool samples were collected before the treatment with NBT-NM108 (Baseline). Three patients from the enrolled patients consumed NBT-NM108 three times a day at 60 g/day for 8 weeks. Two patients further consumed NBT-NM108 for four more weeks (a total of 12 weeks). Stool and blood samples were collected at 3 time points (baseline, 8 weeks post-NBT-NM108, and 12 weeks post-NBT-NM108). We have investigated the effect of NBT-NM108 on gut microbiota and immune parameters involved in MS.

ELIGIBILITY:
Inclusion Criteria:

Patients with the first demyelinating event who meet the McDonald criteria for relapsing remitting MS.

Exclusion Criteria:

1. Primary or secondary progressive MS.
2. Patients with autoimmune comorbidities.
3. Having received prior chemotherapy.
4. Having received Dimethylfumarate (DMF).
5. Pregnant women.
6. Cognitively impaired.
7. Antibiotic use within last 6 months.
8. Probiotic use within 2 months.
9. Self-reported allergy or intolerance to any ingredients in the fiber supplement.
10. Self-reported or diagnosed gastrointestinal symptoms, disorders or adenomas.
11. Active or history of malignant tumors.

Ages: 21 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2022-03-21 (Actual); Primary Completion 2024-06-30 (Actual); Study Completion 2024-07-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Suhayl Dhib-Jalbut, MD, Principal Investigator — Rutgers-RWJMS
Locations (1):
- Robert Wood Johnson University Hospital, New Brunswick, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Baseline data was collected from 7 MS patients enrolled in this study. Three out of seven MS patients consumed NBT-NM108 for 8 weeks. Two out of the three MS patients continued the NBT-NM108 treatment for more 4 weeks (total 12 weeks). Stool and blood samples were collected at 3 time points (baseline, 8 week post-NBT-NM108 , and 12 week post-NBT-NM108 ).
  Baseline: 7, 8 weeks post- NBT-NM108 : 3, 12 weeks post- NBT-NM108 : 2
Groups:
- MS Study Cohort: 7 MS patients enrolled in this study. Three out of seven MS patients consumed NBT-NM108 for 8 weeks. Two out of the three MS patients continued the NBT-NM108 treatment for more 4 weeks (total 12 weeks)
Period: Baseline
Arm/Group | MS Study Cohort
Started | 7
Completed | 7
Not Completed | 0
Period: NBT-NM108 Treatment for 8 Weeks
Arm/Group | MS Study Cohort
Started | 3
Completed | 3
Not Completed | 0
Period: NBT-NM108 Treatment for 12 Weeks
Arm/Group | MS Study Cohort
Started | 2
Completed | 2
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 7 MS patients enrolled in this study. Baseline data was collected from 7 MS patients. Three out of seven MS patients consumed NBT-NM108 for 8 weeks. Two out of the three MS patients continued the NBT-NM108 treatment for more 4 weeks (total 12 weeks)
Groups:
- Study Cohort: 7 MS patients enrolled in this study. Baseline data was collected from 7 MS patients. Three out of seven MS patients consumed NBT-NM108 for 8 weeks. Two out of the three MS patients continued the NBT-NM108 treatment for more 4 weeks (total 12 weeks)
Arm/Group | Study Cohort
Number analyzed (Participants) | 7
Age, Customized [Mean (Standard Deviation); unit: years] | 46.4 (12.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1
  Not Hispanic or Latino | 5
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 3
  White | 2
  More than one race | 0
  Unknown or Not Reported | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7
MS medication at Baseline [Count of Participants; unit: Participants] — This measurement indicate the number of participants using MS medication at the time of recruitment.
  Participants | 2
Treatment naive [Count of Participants; unit: Participants] | 5

OUTCOME MEASURES:

1. Primary Outcome: Assess the Effect of NBT-NM108 on Serum TNF-alpha Levels in MS Patients
Description: TNF-alpha is involved in MS pathology, therefore, we examined the serum level of TNF-alpha by Luminex multiplex assay.
Time Frame: Baseline; and 8 weeks and 12 weeks post-NBT-NM108 treatment.
Population: Three MS patients consumed dietary fiber three times a day at 60 g/day for 8 weeks. Two out of the three MS patients continued NBT-NM108 treatment for more 4 weeks (total12 weeks). Blood samples were collected at 3 time points (baseline, 8 week post-NBT-NM108, and 12 week post-NBT-NM108).
Measure: Mean (Standard Error); unit: pg/ml
Groups:
- Baseline: MS patients who did not consume or before the start of NBT-NM108 treatment.
- NBT-NM108 Treatment for 8 Weeks.: Three MS patients consumed NBT-NM108 three times a day at 60 g/day for 8 weeks.
- NBT-NM108 Treatment for 12 Weeks: Two MS patients further consumed the NBT-NM108 for more 4 weeks (total 12 weeks)
Arm/Group | Baseline | NBT-NM108 Treatment for 8 Weeks. | NBT-NM108 Treatment for 12 Weeks
Number analyzed (Participants) | 3 | 3 | 2
pg/ml | 25.62 (1.28) | 22.58 (0.78) | 20.73 (0.56)

2. Primary Outcome: Examine the Effect of NBT-NM108 on Anaerostipes in MS Patients.
Description: The abundance of the bacteria genus "Anaerostipes" is often found to be decreased in MS patients compared to healthy individuals, indicating a potential link in MS disease progression. Therefore, we examined the abundance by 16s rRNA sequencing of V3-V4 region.
Time Frame: Baseline; and 8 weeks and 12 weeks post-NBT-NM108 treatment.
Population: Baseline data was collected from seven MS patients. Three out of seven MS patients consumed dietary fiber three times a day at 60 g/day for 8 weeks. Two out of the three MS patients continued the HFS treatment for more 4 weeks (total 12 weeks). Stool samples were collected at 3 time points (baseline, 8 week post- NBT-NM108, and 12 week post- NBT-NM108).
Measure: Mean (Standard Error); unit: % abundance
Groups:
- Baseline: This arm includes MS Patients who did not consume NBT-NM108 or MS patients before the start of NBT-NM108 treatment.
- NBT-NM108 Treatment for 8 Weeks: Three MS Patients received NBT-NM108 for 8 weeks. Patients consumed NBT-NM108 three times a day at 60 g/day
- NBT-NM108 Treatment for 12 Weeks: Two MS Patients from arm-2 continued NBT-NM108 for 12 weeks. Patients consumed NBT-NM108 three times a day at 60 g/day
Arm/Group | Baseline | NBT-NM108 Treatment for 8 Weeks | NBT-NM108 Treatment for 12 Weeks
Number analyzed (Participants) | 7 | 3 | 2
% abundance | 1.94 (0.89) | 4.23 (0.52) | 4.52 (0.35)

3. Primary Outcome: Effect of NBT-NM108 on Fecal Lcn-2 Levels in MS Patients
Description: Recently, we found that fecal Lcn-2 level is a sensitive biological indicator for gut dysbiosis in MS. Fecal Lcn-2 levels are increased upon development of gut dysbiosis. Therefore, we measured fecal Lcn-2 levels at baseline, 8 and 12 weeks of HFS treatment.
Time Frame: Baseline, and 8 weeks and 12 weeks post-NBT-NM108 treatment.
Population: as for outcome 2
Measure: Mean (Standard Error); unit: ng/mg
Groups:
- Baseline: This arms includes MS Patients who did not consume NBT-NM108 or MS patients before the start of NBT-NM108 treatment.
  No intervention: MS Patients did not receive NBT-NM108 at 60 g/day.
- NBT-NM108 Treatment for 8 Weeks: Three MS Patients received NBT-NM108 for 8 weeks. Patients consumed dietary fiber three times a day at 60 g/day
- NBT-NM108 Treatment for 12 Weeks: Two MS Patients from arm-2 continued NBT-NM108 for 12 weeks. Patients consumed dietary fiber three times a day at 60 g/day
Arm/Group | Baseline | NBT-NM108 Treatment for 8 Weeks | NBT-NM108 Treatment for 12 Weeks
Number analyzed (Participants) | 7 | 3 | 2
ng/mg | 68.7 (30.9) | 24.4 (3.8) | 33.4 (2.7)

ADVERSE EVENTS:
Time Frame: A nurse from the research team followed up with MS patients by phone at the end of the first week after intervention to check the compliance and adverse effects and then every month thereafter, up to 30 days after the last dose of study intervention. Dr. Suhyal Dhib-Jalbut informed consent to participants and recorded all events from treatment-start date until -end date.
Description: Adverse events were determined based on the FDA guidelines 21CFR312.32.
Groups:
- MS Study Cohort: 7 MS patients enrolled in this study. Baseline data was collected from 7 MS patients. Three out of seven MS patients consumed NBT-NM108 for 8 weeks. Two out of the three MS patients continued the NBT-NM108 treatment for more 4 weeks (total 12 weeks)
Arm/Group | MS Study Cohort
All-Cause Mortality (participants affected / at risk) | 0/7
Serious Adverse Events (participants affected / at risk) | 0/7
Other Adverse Events (participants affected / at risk) | 0/7

LIMITATIONS AND CAVEATS:
We were unable to enroll proposed number of MS patients due to the COVID pandemic.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-08-09): https://cdn.clinicaltrials.gov/large-docs/24/NCT04574024/Prot_SAP_002.pdf
  • Informed Consent Form (2023-03-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT04574024/ICF_001.pdf